CLINICAL TRIAL: NCT00004936
Title: Role of Radiology in the Pretreatment Evaluation of Invasive Cervical Cancer
Brief Title: MRI and CT Scans to Evaluate Invasive Cervical Cancer Before Treating Patients
Acronym: ACRIN 6651
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Diagnostic
Other Study IDs: CDR0000067622; ACRIN-6651; GOG-183; CA80098 (Other Grant/Funding Number: NCI CIP)
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Cervical Cancer
Keywords: stage III cervical cancer; stage IB cervical cancer; stage IIB cervical cancer; stage IVB cervical cancer; stage IIA cervical cancer; stage IVA cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma; cervical adenosquamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Magnetic Resonance Spectroscopy; Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: iodinated contrast dye
Procedure: computed tomography
Procedure: magnetic resonance imaging
Radiation: gadopentetate dimeglumine

SUMMARY:
RATIONALE: Imaging procedures such as MRI or CT scans may improve the ability to detect cervical cancer and determine the extent of disease.

PURPOSE: Diagnostic trial to determine the effectiveness of MRI and CT scans in evaluating invasive cervical cancer before treatment of patients.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the diagnostic performance of magnetic resonance imaging (MRI), computed tomography (CT), and clinical FIGO staging in patients with invasive cervical cancer.
* Compare the accuracy of MRI, CT, and clinical FIGO staging in the evaluation of morphologic tumor prognostic factors in FIGO stage IB1 and stage IB2 and greater in these patients.
* Examine the value of imaging assessment of tumor prognostic factors (alone or in combination) as predictors of recurrence within 2 years of surgery in these patients.
* Evaluate the quality of life in the 12-month period after staging and treatment to potentially change staging accuracy.

OUTLINE: This is a multicenter study.

Patients undergo a computed tomography scan with iodinated contrast dye followed by a magnetic resonance imaging scan with or without contrast comprising gadopentetate dimeglumine or vice versa.

Within 6 weeks of first protocol imaging study, patients undergo one of the following surgeries:

* Laparoscopic, transabdominal, or transvaginal hysterectomy
* Extrafascial total abdominal hysterectomy
* Trachelectomy Quality of life is assessed at 1 and 12 months.

Patients are followed every 3 months for 1 year and then every 6 months for 1 year.

PROJECTED ACCRUAL: A total of 465 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive cervical cancer, including invasive squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma

  * FIGO stage IB1 with clinically visible gross lesion OR
  * FIGO stage IB2 or greater
* Scheduled for one of the following surgeries at a participating Gynecological Oncology Group center:

  * Laparoscopic, transabdominal, or transvaginal hysterectomy
  * Extrafascial total abdominal hysterectomy
  * Trachelectomy
* Not scheduled for a loop electrosurgical excision procedure or a cone biopsy only

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* No cardiac pacemakers

Pulmonary:

* No asthma

Other:

* Not pregnant
* No contraindication to computed tomography (CT) (e.g., history of allergy to CT contrast medium)
* No contraindication to magnetic resonance imaging (e.g., intracranial vascular clip)
* No nonmalignant general medical or psychiatric condition that would preclude consent or surgery

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for invasive cervical cancer

Surgery:

* See Disease Characteristics
* No prior surgery for invasive cervical cancer

Other:

* No prior medical treatment for invasive cervical cancer

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-04; Primary Completion 2001-05 (Actual); Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hedvig Hricak, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York

REFERENCES:
- [Result] Mitchell DG, Snyder B, Coakley F, Reinhold C, Thomas G, Amendola MA, Schwartz LH, Woodward P, Pannu H, Atri M, Hricak H. Early invasive cervical cancer: MRI and CT predictors of lymphatic metastases in the ACRIN 6651/GOG 183 intergroup study. Gynecol Oncol. 2009 Jan;112(1):95-103. doi: 10.1016/j.ygyno.2008.10.005. Epub 2008 Nov 20. PMID 19019414
- [Result] Hricak H, Gatsonis C, Coakley FV, Snyder B, Reinhold C, Schwartz LH, Woodward PJ, Pannu HK, Amendola M, Mitchell DG. Early invasive cervical cancer: CT and MR imaging in preoperative evaluation - ACRIN/GOG comparative study of diagnostic performance and interobserver variability. Radiology. 2007 Nov;245(2):491-8. doi: 10.1148/radiol.2452061983. PMID 17940305
- [Result] Mitchell DG, Snyder B, Coakley F, Reinhold C, Thomas G, Amendola M, Schwartz LH, Woodward P, Pannu H, Hricak H. Early invasive cervical cancer: tumor delineation by magnetic resonance imaging, computed tomography, and clinical examination, verified by pathologic results, in the ACRIN 6651/GOG 183 Intergroup Study. J Clin Oncol. 2006 Dec 20;24(36):5687-94. doi: 10.1200/JCO.2006.07.4799. PMID 17179104
- [Result] Amendola MA, Hricak H, Mitchell DG, Snyder B, Chi DS, Long HJ 3rd, Fiorica JV, Gatsonis C. Utilization of diagnostic studies in the pretreatment evaluation of invasive cervical cancer in the United States: results of intergroup protocol ACRIN 6651/GOG 183. J Clin Oncol. 2005 Oct 20;23(30):7454-9. doi: 10.1200/JCO.2004.00.5397. PMID 16234512
- [Result] Hricak H, Gatsonis C, Chi DS, Amendola MA, Brandt K, Schwartz LH, Koelliker S, Siegelman ES, Brown JJ, McGhee RB Jr, Iyer R, Vitellas KM, Snyder B, Long HJ 3rd, Fiorica JV, Mitchell DG; American College of Radiology Imaging Network 6651; Gynecologic Oncology Group 183. Role of imaging in pretreatment evaluation of early invasive cervical cancer: results of the intergroup study American College of Radiology Imaging Network 6651-Gynecologic Oncology Group 183. J Clin Oncol. 2005 Dec 20;23(36):9329-37. doi: 10.1200/JCO.2005.02.0354. PMID 16361632